CLINICAL TRIAL: NCT04275921
Title: Magnetic Resonance Imaging for Lung Radiotherapy a Prospective Study
Brief Title: Magnetic Resonance Imaging for Lung Radiotherapy
Acronym: MRI Lung
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Clatterbridge Cancer Centre NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CO996
Record Dates: First submitted 2020-02-11; First posted 2020-02-19 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-02

CONDITIONS: Cancer; Lung Cancer
Keywords: MRI; Radiotherapy
MeSH Terms: conditions — Neoplasms; Lung Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study participants cohort I (Experimental): 3 stage III NSCLC patients receiving radiotherapy will be imaged, each for a single MRI session using TWIST and HASTE sequences.
  Interventions: Diagnostic Test: MRI scan; Diagnostic Test: 4D MRI
- Study participants cohort II (Experimental): 12 patients will be imaged, each for two MRI sessions taking place during the radiotherapy schedule and separated by at least a week.
  Interventions: Diagnostic Test: MRI scan; Diagnostic Test: 4D MRI

INTERVENTIONS:
Diagnostic Test: MRI scan — MRI analysis using TWIST and HASTE
Diagnostic Test: 4D MRI — 4D MRI alongside 4D CT in lung cancer

SUMMARY:
The purpose of this study is to investigate the use of Magnetic Resonance Imaging (MRI) in the diagnostic and planning phase of radiotherapy for lung cancer and then introduce it into on-treatment imaging to improve the accuracy of radiotherapy. The study compromises of two phases, a technical phase followed by a clinical phase.

The aim of the technical phase is to develop and test MR sequences using a diagnostic scanner for use in the chest.

This will be carried out on a humanoid phantom and subsequently healthy volunteers.

The second phase will be a clinical phase to assess the accuracy of visualising all thoracic structures and the tumour in lung cancer patients using the defined MR sequences. It will compromise of 2 parts; the first part will involve 3 lung cancer patients as a pilot to enable the fine tuning of the sequences. The 2nd part will involve the evaluation of MRI in relation to planning CT in 12 lung cancer patients.

The hypothesis is that the use of 4D MRI will be more accurate in defining the tumour and intrathoracic structures thanachieved with the current standard of 4DCT to improve the accuracy and potentially the outcome of radical radiotherapy for non-small cell lung cancer.

DETAILED DESCRIPTION:
Firstly, 3 stage III NSCLC patients receiving radiotherapy will be imaged, each for a single MRI session using TWIST and HASTE sequences. Initial sequence parameters will be those determined during the preceding technical development, but these will be fine-tuned to maximize tumour visualisation as this part of the study progresses, achieving the most practically useful trade-off between image resolution and noise, qualitatively and quantitatively assessed by a radiologist to determine and fine-tune image quality.

Then a further 12 patients will be imaged, each for two MRI sessions taking place during the radiotherapy schedule and separated by at least a week. Each MR session will consist of the following sequence: 15 seconds of TWIST, 15 seconds of HASTE, 90 seconds off, 15 seconds of TWIST and 15 seconds of HASTE. For each patient an on-treatment 4D cone-beam CT will also be collected (standard process), alongside the diagnostic quality planning 4DCT. Patient breathing coaching will be consistent between CT and MR, as will patient positioning; that is, patients will be imaged with their arms above their heads. The images will be analyzed to determine -

1. Do extents of tumour movement seen in TWIST 4D-MR images differ from those seen in planning 4D-CT scans, judging the movement extent according to differences in internal target and gross tumour volumes (ITVs and GTVs) defined from the two sets of images, and in the range of motion of the tumour centre of mass? This may well be the case, since the 4D-MR scans catalogue movement over several breathing cycles, whereas 4D-CTs describe a single composite cycle, synthesised from slices collected at various times over multiple cycles.
2. How reproducible is the movement seen at the two MR imaging sessions? Additionally, how reproducible is the movement seen within each MR imaging session?
3. How similar according to volume, Dice similarity index (percentage of overlap) and Haussdorf distance (maximum distance between the contours of two structures) are GTVs outlined on single phases of 4D-CT and TWIST 4D-MR images, after rigidly registering the centres-of-mass of the two GTVs to allow for movement?
4. How consonant are tumour contours defined on single slice HASTE MR images with those defined on a phase of the 4D TWIST images? Answering question 1 will allow us to determine the utility of gauging tumour movement over extended 4D-MR imaging sessions, rather than from 4D-CT sessions which have to be short to avoid excessively irradiating patients. Question 2 will cast further light on the same issue, allowing us to determine the stability over the course of RT schedules of motion assessed over the course of around 1 minute during an individual TWIST scan.

Answering question 3 will allow us to understand how fully 4D-MR images can be used within the treatment planning process. If outlined GTVs differ greatly between MRI and CT, then 4D-MRI might only provide more complete movement data; whereas if CT and MRI-based GTVs are similar the 4D-MRI may have more uses in treatment planning, particularly if some tumour regions are more clearly visible on MRI than on CT.

Question 4 will allow us to gauge the accuracy and precision of tumour definition on real-time single MRI slices, compared to definition on 4D-MR and 4D-CT. Answering this question is an essential precursor to the development of automatic algorithms

ELIGIBILITY:
Inclusion Criteria:

This study will recruit patients due to have radical external beam radiotherapy as per standard institutional practice.

The criteria specified in the institutional protocol are:

* Histologically verified NSCLC or presumed not histologically verified but MDT reviewed and agreed if obtaining biopsy is considered too risky
* Stage II, IIIA & IIIB (AJCC, 7th Edition TNM), fully staged with CT, PET-CT +/-EBUS for mediastinal staging
* WHO performance status ≤ 2
* Adequate respiratory function
* Absence of malignant effusion
* Aged 18 and over

Exclusion Criteria:

* Under 18 years or age
* Patients not able to have radical radiotherapy
* Pregnant or lactating women
* Unable to give informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-05-16 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
The aim of the technical phase is to develop and test MR sequences using a diagnostic scanner for use in the chest | 2 years
  Measure gross tumour volume (Gross Tumour Volume/ tumour) and normal structures. Two clinical oncologists are generate consensus based tumour motion envelopes on image datasets comprising anatomical planes oriented along each cardinal axis. Dice similarity index (percentage of overlap) and Haussdorf distance (maximum distance between the contours of two structures) are gross tumour volumes s outlined on single phases of 4D-CT and TWIST 4D-MR images, after rigidly registering the centres-of-mass of the two gross tumour volumes.

SECONDARY OUTCOMES:
4D MRI will be compared to 4D CT as an imaging methodology | 2 years
  Image outlines are merged to create a single representation of the tumour surface comparable or better than 4D-CT. This merged tumour surface will be compared to the standard 4D-CT tumour outline using Haussdorf and Dice metrics. An anthropomorphic phantom will also be 4D-CT and 4D-MR imaged and outlined, providing ground-truth data with which to determine the relative accuracies of CT and MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Brada, PhD, MD, Principal Investigator — Clatterbridge Cancer Centre
Locations (1):
- Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, United Kingdom

IPD SHARING:
Plan to Share IPD: No